CLINICAL TRIAL: NCT00981500
Title: Effect of Bariatric Surgery-induced Weight Loss on Glucose Homeostasis
Brief Title: Glucose Homeostasis Pre and Post Bariatric Surgery
Acronym: RB
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-0175
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Morbid Obesity
Keywords: obesity; gastric bypass; gastric banding; weight loss; insulin sensitivity; sleeve gastrectomy; fibroblast growth factor 21; fibroblast growth factor 19
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss; Insulin Resistance | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, tongue tissue, muscle tissue, fat tissue,liver tissue, colon tissue, stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Gastric Bypass: morbidly obese subjects undergoing gastric bypass surgery
  Interventions: Procedure: gastric bypass
- gastric banding: morbidly obese subjects undergoing laparoscopic gastric banding surgery
  Interventions: Procedure: gastric banding
- sleeve gastrectomy: morbidly obese subjects undergoing sleeve gastrectomy
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: gastric bypass — Roux-en-Y gastric bypass
  Other Names: Roux-en-Y gastric bypass
  Groups: Gastric Bypass
Procedure: gastric banding — laparoscopic adjustable gastric banding
  Other Names: lap band
  Groups: gastric banding
Procedure: sleeve gastrectomy — vertical sleeve gastrectomy
  Other Names: gastric sleeve
  Groups: sleeve gastrectomy

SUMMARY:
The investigators wish to study the effects of three forms of bariatric surgery: Roux-en-Y gastric bypass, Sleeve Gastrectomy, and Gastric Banding. The surgery is not part of the clinical trial. If your insurance does not cover the procedure, then you are responsible for payment of the surgical process. We are doing pre and post surgery testing to provide a better understanding of the effect of bariatric surgery-induced weight loss on metabolic function.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective weight loss therapy for obesity. Moreover, the early improvement in insulin sensitivity and the resolution of type 2 diabetes after bariatric surgery has led to the hypothesis that bariatric surgery has specific beneficial effects on glucose homeostasis beyond weight loss alone. However, this hypothesis has never been adequately evaluated in human subjects. Therefore, the primary goal of this proposal is to provide a better understanding of the effect of bariatric surgery-induced weight loss on insulin action and pancreatic beta cell function.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m²
* on stable dose of medications for at least 4 weeks before the pre-surgery metabolic studies

Exclusion Criteria:

* smokes > 7 cigarettes per day
* previous malabsorptive or restrictive intestinal surgery
* pregnant or breastfeeding
* recent history of neoplasia (< 5 years ago)
* have malabsorptive syndromes and inflammatory intestinal disease
* diabetes mellitus
* show signs of oral disease or xerostomia (i.e., dry mouth)
* history of chronic rhinitis
* on medication that might affect metabolism
* severe organ dysfunction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 (per surgical group) morbidly obese (BMI ≥ 35 kg/m²) subjects scheduled for bariatric surgical procedures will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The effect of bariatric surgery-induced weight loss (Roux-en-Y gastric bypass, sleeve gastrectomy, and laparoscopic adjustable banding) on insulin action | at 20% weight loss post surgery

SECONDARY OUTCOMES:
The effect of bariatric surgery-induced weight loss Roux-en-Y gastric bypass, sleeve gastrectomy, and laparoscopic adjustable gastric banding) on pancreatic beta cell response | at 20% weight loss post surgery
Determine the effect of bariatric surgery induced weight loss (Roux-en-Y gastric bypass, sleeve gastrectomy, and laparoscopic adjustable gastric banding) on gut microbiota. | at 20% weight loss post surgery
Identify host genes that co-vary with an altered metagenome in obese individuals that undergo bariatric surgery | at 20% weight loss post surgery.
Investigate how the metagenome is affected by bariatric surgery procedures leading to weight reduction | at 20% weight loss post surgery
The effect of bariatric surgery-induced weight loss (Roux-en-Y gastric bypass, sleeve gastrectomy, and laparoscopic adjustable gastric banding) on postprandial plasma fibroblast growth factor (FGF)21 and FGF19 responses. | at 20% weight loss post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoshino J, Patterson BW, Klein S. Adipose Tissue CTGF Expression is Associated with Adiposity and Insulin Resistance in Humans. Obesity (Silver Spring). 2019 Jun;27(6):957-962. doi: 10.1002/oby.22463. Epub 2019 Apr 19. PMID 31004409
- [Derived] Harris LLS, Smith GI, Mittendorfer B, Eagon JC, Okunade AL, Patterson BW, Klein S. Roux-en-Y Gastric Bypass Surgery Has Unique Effects on Postprandial FGF21 but Not FGF19 Secretion. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3858-3864. doi: 10.1210/jc.2017-01295. PMID 28938478
- [Derived] Magkos F, Bradley D, Eagon JC, Patterson BW, Klein S. Effect of Roux-en-Y gastric bypass and laparoscopic adjustable gastric banding on gastrointestinal metabolism of ingested glucose. Am J Clin Nutr. 2016 Jan;103(1):61-5. doi: 10.3945/ajcn.115.116111. Epub 2015 Nov 25. PMID 26607940
- [Derived] Bradley D, Magkos F, Eagon JC, Varela JE, Gastaldelli A, Okunade AL, Patterson BW, Klein S. Matched weight loss induced by sleeve gastrectomy or gastric bypass similarly improves metabolic function in obese subjects. Obesity (Silver Spring). 2014 Sep;22(9):2026-31. doi: 10.1002/oby.20803. Epub 2014 May 28. PMID 24891156
- [Derived] Magkos F, Bradley D, Schweitzer GG, Finck BN, Eagon JC, Ilkayeva O, Newgard CB, Klein S. Effect of Roux-en-Y gastric bypass and laparoscopic adjustable gastric banding on branched-chain amino acid metabolism. Diabetes. 2013 Aug;62(8):2757-61. doi: 10.2337/db13-0185. Epub 2013 Apr 22. PMID 23610059
- [Derived] Kohli R, Bradley D, Setchell KD, Eagon JC, Abumrad N, Klein S. Weight loss induced by Roux-en-Y gastric bypass but not laparoscopic adjustable gastric banding increases circulating bile acids. J Clin Endocrinol Metab. 2013 Apr;98(4):E708-12. doi: 10.1210/jc.2012-3736. Epub 2013 Mar 1. PMID 23457410